CLINICAL TRIAL: NCT00837655
Title: Study of the Effect of Treatment With Sevelamer on Glucose Tolerance and Insulin Sensitivity in Patients With Chronic Renal Failure
Brief Title: Effect of Sevelamer on Glucose Tolerance and Insulin Sensitivity in Patients With Chronic Renal Failure (CKD)
Acronym: SIR
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI retired
Sponsor: Karolinska Institutet (Other)
Collaborators: Göteborg University (Other)
Responsible Party: Anders Alvestrand, Professor, Karolinska institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SIR_CT_CLINTEC_01
Record Dates: First submitted 2009-01-29; First posted 2009-02-05 (Estimated); Last update posted 2012-09-26 (Estimated); Status verified 2009-01

CONDITIONS: Kidney Failure, Chronic; End-Stage Renal Disease; Insulin Resistance; Hyperphosphatemia
Keywords: Chronic kidney disease; End-stage renal disease; phosphate binder; insulin resistance; glucose intolerance; sevelamer
MeSH Terms: conditions — Kidney Failure, Chronic; Insulin Resistance; Hyperphosphatemia; Renal Insufficiency, Chronic; Glucose Intolerance | interventions — Sevelamer; Calcium Carbonate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Sevelamer intervention
  Interventions: Drug: Sevelamer
- 2 (Active Comparator): Calcium carbonate
  Interventions: Drug: Calcium carbonate

INTERVENTIONS:
Drug: Sevelamer — sevelamer tablets, 800 mg (Renagel(r), Genzyme Inc). The initial daily dose of sevelamer will be 2400 mg (800 mg x 3). After the first week of treatment the dose will be increased to 4800 mg. If treatment with sevelamer is well tolerated and if a phosphate concentration of <1.8 mmol/l is not obtained, the dose may be increased further. The maximum daily dose of sevelamer will be 9600 mg. If a patient experiences side effects, the dose of sevelamer will be reduced to the highest acceptable dose, and, if a phosphate concentration of <1.8 mmol/l is not obtained, the treatment will be supplemented with calcium carbonate in a dose tolerated by the patient.
  Other Names: Renagel
  Arms: 1
Drug: Calcium carbonate — Calcium carbonate tablets, 250 mg (Kalcidon, Abigo AB). Calcium carbonate will be prescribed at the dose given prior to the washout period. The dose will be adjusted weekly to obtain a serum phosphate concentration <1.8 mmol/l.
  Arms: 2

SUMMARY:
The purpose of this study is to perform a randomized, controlled clinical trial to investigate if the phosphate binder sevelamer can improve insulin resistance and glucose handling in patients receiving maintenance hemodialysis.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients 18-80 years of age with chronic renal failure treated with maintenance HD for >3 months.

Exclusion Criteria:

* Diabetes mellitus
* Treatment with sevelamer within 3 months prior to enrollment
* Acute, clinically significant inflammation within 1 month prior to enrollment
* Pregnancy or breast-feeding
* Clinically significant obstipation or bowel obstruction
* Discontinuation of previous sevelamer treatment because of side effects
* Expected time in HD < 1 year
* Unwillingness to undergo the investigations and follow-up required in the the protocol
* Patients who have received any investigational drug within 1 month prior to enrolment
* Participation in another study, which may interfere with the present study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-01; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Change in insulin sensitivity and/or glucose tolerance from baseline to the end of the study, as obtained by ISIOGTT. | Week 12

SECONDARY OUTCOMES:
Change from baseline to the end of the trial in surrogate markers of phosphate balance (PTH, s-urea, s-creatinine, ionized Ca, phosphate). | Week 12
Change from baseline to end of the study in markers of lipid homeostasis (total cholesterol, LDL, HDL, ApoA, ApoB, TG, free fatty acids) | Week 12
Change from baseline to the end of the study in circulating inflammatory cytokines (hsCRP, TNF, fibrinogen, PAI, fetuin) | Week 12
Number of adverse events directly attributable to sevelamer or calciumcarbonate treatments. | Weekly until end of study

CONTACTS AND LOCATIONS:
Overall Officials: Anders Alvestrand, MD PhD, Principal Investigator — Karolinska Institutet; Jonas Axelsson, MD, PhD, Principal Investigator — Karolinska Institutet
Locations (2):
- Sweden (2):
  - Sahlgrenska University Hospital, Gothenburg, Gothenburg
  - Karolinska University Hospital, Stockholm, Stockholm County

REFERENCES:
- [Background] Soonthornpun S, Setasuban W, Thamprasit A, Chayanunnukul W, Rattarasarn C, Geater A. Novel insulin sensitivity index derived from oral glucose tolerance test. J Clin Endocrinol Metab. 2003 Mar;88(3):1019-23. doi: 10.1210/jc.2002-021127. PMID 12629079